CLINICAL TRIAL: NCT07007884
Title: The Effect of Transauricular Vagal Nerve Stimulation (taVNS) on Cardiac Autonomic Functions in Patients With Spinal Cord Injury
Brief Title: Effect of Transauricular Vagal Stimulation on Cardiac Function After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayşenur ŞİMŞEK YAĞLIOĞLU, medical doctor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: E2-23-3620
Record Dates: First submitted 2025-05-21; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injury (SCI)
Keywords: vagus nerve stimülation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Patients were divided into groups as group I cervical complete spinal cord injury (SCI) patients in active transauricular vagal nerve stimülation (taVNS) group, group II cervical complete SCI patients in sham taVNS group and group III lumbar SCI patients (diagnosed with cauda equina syndrome) in active taVNS group.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cervical spinal cord injury - Active taVNS (Experimental): The study included 30 traumatic spinal cord injury (SCI) patients who fulfilled the criteria. Patients were divided into groups as group I cervical complete SCI patients in active transaurikular vagal nerve stimülation (taVNS) group (n:10), group II cervical complete SCI patients in sham taVNS group (n:10) and group III lumbar SCI patients (diagnosed with cauda equina syndrome) in active taVNS group (n:10).
  Interventions: Device: Active Transauricular Vagus Nerve Stimulation
- Cervical spinal cord injury - Sham taVNS (Experimental): The study included 30 traumatic SCI patients who fulfilled the criteria. Patients were divided into groups as group I cervical complete SCI patients in active taVNS group (n:10), group II cervical complete SCI patients in sham taVNS group (n:10) and group III lumbar SCI patients (diagnosed with cauda equina syndrome) in active taVNS group (n:10).
  Interventions: Device: Sham Transauricular Vagus Nerve Stimulation
- Lumbar spinal cord injury (Cauda Equina Syndrome)- Active taVNS (Experimental): The study included 30 traumatic spinal cord injury (SCI) patients who fulfilled the criteria. Patients were divided into groups as group I cervical complete SCI patients in active taVNS group (n:10), group II cervical complete SCI patients in sham taVNS group (n:10) and group III lumbar SCI patients (diagnosed with cauda equina syndrome) in active taVNS group (n:10).
  Interventions: Device: Active Transauricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Active Transauricular Vagus Nerve Stimulation — Active taVNS application was performed by stimulating a sterile acupuncture needle (0.25x25 mm) placed on the left ear cymba choncae with a stimulator. Active taVNS group received for 10 days, 30 minutes with a current intensity of 1 mA, pulse width of 200 µs, frequency of 25 Hz and biphasic sinusoidal waveform. In the sham group, stimulation was applied to the lobulus auriculae of the left ear (which is not innervated by the vagus nerve) using the same current intensity and duration as the active group.
  Other Names: taVNS, auricular VNS
  Arms: Cervical spinal cord injury - Active taVNS; Lumbar spinal cord injury (Cauda Equina Syndrome)- Active taVNS
Device: Sham Transauricular Vagus Nerve Stimulation — Sham taVNS application was performed by stimulating a sterile acupuncture needle (0.25x25 mm) placed on the left lobulus auriculae of the left ear (which is not innervated by the vagus nerve) with a stimulator. Sham taVNS group received for 10 days, 30 minutes with a current intensity of 1 mA, pulse width of 200 µs, frequency of 25 Hz and biphasic sinusoidal waveform.
  Arms: Cervical spinal cord injury - Sham taVNS

SUMMARY:
The aim of this study is to investigate the effect of transauricular vagal nerve stimulation (taVNS) on cardiac autonomic functions in patients with spinal cord injury (SCI).

DETAILED DESCRIPTION:
Spinal cord injury impairs autonomic pathways and ultimately cardiovascular homeostasis. Spinal cord injury affects the autonomic system, resulting in impaired cardiac autonomic functions. This study is designed to evaluate the effect of transauricular vagal nerve stimulation (taVNS) on cardiac autonomic functions in patients with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18-60
2. Having a traumatic spinal cord injury
3. Cervical spinal cord injury patients with a history of autonomic dysreflexia
4. At least 6 months after the injury
5. Signing an informed consent form showing consent to participate in the study

Exclusion Criteria:

1. Having a cardiac or neural pacemaker
2. Presence of pregnancy
3. Clinical coronary artery disease confirmed by invasive or coronary computed tomographic angiography
4. History of acute coronary syndrome (unstable angina, myocardial infarction)
5. Documented arrhythmia and/or use of antiarrhythmic drugs on ECG
6. Diagnosis of hypertension and use of antihypertensive drugs
7. Damaged skin lesion in the application area

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-07-16 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Low frequency/ High frequency (LF/HF) | At baseline (Day 0), Day 1, Day 10, and Day 11
  Heart rate variability (HRV) is considered an indicator of neural control over the heart and is measured by analyzing the variations in NN intervals between consecutive R waves on an electrocardiogram (ECG).Frequency-domain analyses determine the power of fluctuations in heart rate signals within specific frequency bands. This analysis can be conducted using short-term Holter ECG recordings or data from 5-minute segments of a 24-hour Holter ECG. In our study, the short-term effects of taVNS on frequency domain HRV parameters will be evaluated using data obtained from 24-hour Holter ECG recordings on the pre-stimulation day (day 0) and day 11, and the acute effects will be assessed using data from 15-minute Holter recordings on day 1 and day 10.The LF/HF ratio is also one of the frequency-domain HRV parameters.
  LF/HF (ratio): low-to-high frequency power ratio The LF/HF ratio serves as an indicator of sympathovagal balance.

SECONDARY OUTCOMES:
Total Power | At baseline (Day 0) and Day 11
  Frequency-domain heart rate variability (HRV) parameters include Total Power, Ultra Low Frequency (ULF), Very Low Frequency (VLF), Low Frequency (LF), High Frequency (HF), and the Low Frequency/High Frequency (LF/HF) ratio.
  Total power, represents the total power of all frequency components within the frequency spectrum. It is the sum of the very low frequency (VLF), low frequency (LF), and high frequency (HF) components. Total power is an important parameter for the overall evaluation of autonomic nervous system functions.
  In our study, the short-term effects of taVNS on total power will be evaluated using data obtained from 24-hour Holter ECG recordings on the pre-stimulation day (day 0) and on day 11.
  Total power (millisecond²: ms²): Variance of all NN(Normal-to-Normal) intervals (<0.4 Hz)
Ultra Low Frequency (ULF) | At baseline (Day 0) and Day 11
  The ULF is also one of the frequency-domain HRV parameters. ULF represents the ultra low frequency. It indicates frequencies <0.003 Hz. It does not directly reflect sympathetic or parasympathetic activity.
  In our study, the short-term effects of taVNS on ULF will be evaluated using data obtained from 24-hour Holter ECG recordings on the pre-stimulation day (day 0) and on day 11.
  ULF (ms²): ultra low frequency (<0.003 Hz)
Very Low Frequency (VLF) | At baseline (Day 0) and Day 11
  The VLF is also one of the frequency-domain HRV parameters. VLF represents the very low frequency. It indicates frequencies between <0.003 and 0.04 Hz. It has been associated with baroreceptor activity, thermoregulation, the renin-angiotensin system, and endothelial functions.
  In our study, the short-term effects of taVNS on VLF will be evaluated using data obtained from 24-hour Holter ECG recordings on the pre-stimulation day (day 0) and on day 11.
  VLF (ms²): very low frequency (frequencies between <0.003 and 0.04 Hz)
Low Frequency (LF) | At baseline (Day 0), Day 1, Day 10, and Day 11
  The LF is also one of the frequency-domain HRV parameters. LF represents the low frequency. It indicates frequencies between 0.04 and 0.15 Hz. It reflects a combination of sympathetic and parasympathetic activity and is particularly associated with sympathetic activity in seated or standing positions.
  In our study, the short-term effects of taVNS on LF will be evaluated using data obtained from 24-hour Holter ECG recordings on the pre-stimulation day (day 0) and on day 11, while the acute effects will be assessed using data from 15-minute Holter recordings on day 1 and day 10.
  LF (ms2): low frequency power (0.04 to 0.15)
High Frequency (HF) | At baseline (Day 0), Day 1, Day 10, and Day 11
  The HF is also one of the frequency-domain HRV parameters. HF represents the high frequency. It indicates frequencies between 0.15 and 0.40 Hz. It reflects parasympathetic activity. An increase in HF indicates a high vagal tone.
  In our study, the short-term effects of taVNS on HF will be evaluated using data obtained from 24-hour Holter ECG recordings on the pre-stimulation day (day 0) and on day 11, while the acute effects will be assessed using data from 15-minute Holter recordings on day 1 and day 10.
  HF (ms²): high frequency power (0.15 to 0.40)
SDNN: Standard Deviation of NN intervals | At baseline (Day 0) and Day 11
  Time-domain HRV parameters are based on the analysis of the time intervals between normal heartbeats in 24-hour ECG recordings. In our study, the time-domain HRV parameters, including SDNN, SDNNi, SDANN, RMSSD, and pNN50, will be calculated from 24-hour Holter ECG recordings obtained before stimulation and after 10 days of stimulation.
  SDNN (ms): It is the standard deviation of all NN (interval between two adjacent R waves) intervals in the 24-hour ECG recording.
SDNNi: Mean of the standard deviations of all NN intervals for all 5-minute segments | At baseline (Day 0) and Day 11
  Time-domain HRV parameters are based on the analysis of the time intervals between normal heartbeats in 24-hour ECG recordings. In our study, the time-domain HRV parameters, including SDNN, SDNNi, SDANN, RMSSD, and pNN50, will be calculated from 24-hour Holter ECG recordings obtained before stimulation and after 10 days of stimulation.
  SDNN index (ms): It is the mean of the standard deviations of all NN intervals for all 5-minute segments within 24 hours.
SDANN: Standard deviation of the averages of NN intervals in all 5-minute segments | At baseline (Day 0) and Day 11
  Time-domain HRV parameters are based on the analysis of the time intervals between normal heartbeats in 24-hour ECG recordings. In our study, the time-domain HRV parameters, including SDNN, SDNNi, SDANN, RMSSD, and pNN50, will be calculated from 24-hour Holter ECG recordings obtained before stimulation and after 10 days of stimulation.
  SDANN (ms): The standard deviation of the mean of the normal RR intervals of the 5-minute segments in the 24-hour ECG recording.
RMSSD: Root Mean Square of the Successive Differences | At baseline (Day 0) and Day 11
  Time-domain HRV parameters are based on the analysis of the time intervals between normal heartbeats in 24-hour ECG recordings. In our study, the time-domain HRV parameters, including SDNN, SDNNi, SDANN, RMSSD, and pNN50, will be calculated from 24-hour Holter ECG recordings obtained before stimulation and after 10 days of stimulation.
  RMSDD (ms): is the root of the mean of squares of consecutive NN interval differences over the 24-hour recording.
pNN50: Percentage of successive NN intervals that differ by more than 50 ms | At baseline (Day 0) and Day 11
  Time-domain HRV parameters are based on the analysis of the time intervals between normal heartbeats in 24-hour ECG recordings. In our study, the time-domain HRV parameters, including SDNN, SDNNi, SDANN, RMSSD, and pNN50, will be calculated from 24-hour Holter ECG recordings obtained before stimulation and after 10 days of stimulation.
  pNN50 (%): The proportion of differences between consecutive NN intervals greater than 50 ms during the 24-hour recording
Heart rate response to the tilt test | At baseline (Day 0) and Day 11
  The Ewing's battery parameters (EBP) are the most popular among clinical autonomic test batteries. In our study, the tilt test, heart rate and blood pressure changes, respiratory heart rate changes, and the Valsalva maneuver selected from the EBP clinical autonomic tests.
  This test is used to evaluate the hemodynamic response to changes in body position. When moving from a supine to an upright position, venous pooling in the lower extremities leads to a decrease in stroke volume, resulting in a rapid increase in heart rate within the first 30 seconds. The normal response is characterized by a slight increase in heart rate (by 5-20 beats per minute), and the 30/15 ratio in the test is used to assess the initial phase of adaptation to standing. After tilting to an 80-degree upright position using a tilt table, the ratio of the longest R-R interval around the 30th beat to the shortest R-R interval around the 15th beat is calculated. A ratio lower than 1.04 is considered abnormal.
Blood pressure response to the tilt test | At baseline (Day 0) and Day 11
  It is another of the clinical autonomic tests in our study. This is another test used to evaluate the hemodynamic response to changes in body position. When moving from a supine to an upright position, blood moves to the lower extremities, reducing venous return and stroke volume. This test is performed to identify the presence of orthostatic hypotension (OH). After measuring the patient's baseline blood pressure in the supine position, the patient is brought to an 80-degree upright position using a tilt table and is kept in this position for 5 minutes. A decrease in systolic blood pressure by ≥20 mmHg or in diastolic blood pressure by ≥10 mmHg is considered a positive test result.
Heart rate response to the Valsalva maneuver (Valsalva ratio) | At baseline (Day 0) and Day 11
  It is another of the clinical autonomic tests in our study. The Valsalva maneuver is a test used to evaluate baroreceptor function and reflects parasympathetic activity. In this test, the patient lies in a supine position with the head elevated to 30 degrees, takes a deep breath, and then performs a forced expiration against a closed airway for 15 seconds, followed by a 45-second rest period of normal breathing. The ratio of the longest R-R interval to the shortest R-R interval is recorded. Three maneuvers are performed, and the average of the three ratios is calculated. A value below 1.2 indicates parasympathetic dysfunction.
Respiratory heart rate variability | At baseline (Day 0) and Day 11
  It is another of the clinical autonomic tests in our study. This test is based on the phenomenon of respiratory sinus arrhythmia, which becomes particularly evident when breathing at a rate of six breaths per minute. The test is used to assess the effect of the parasympathetic nervous system on heart rate. In this test, the patient lies in a supine position with the head elevated to 30 degrees and is instructed to breathe in and out six times over one minute, with a 5-second inspiration and a 5-second expiration cycle. The difference between the maximum and minimum heart rate within the one-minute cycle is measured. The cycle is repeated three times, and the average of the heart rate differences is calculated. A variability of less than 10 beats per minute indicates parasympathetic dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ Gaziler Fizik Tedavi ve Rehabilitasyon Eğitim ve Araştırma Hastanesi, Ankara, Turkey (Türkiye)